CLINICAL TRIAL: NCT06268600
Title: The Protection of Thyroid Function in IMRT for Nasopharyngeal Carcinoma: A Retrospective Study
Brief Title: The Protection of Thyroid Function in IMRT for Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NPC-Thyroid function
Record Dates: First submitted 2024-02-13; First posted 2024-02-20 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Nasopharyngeal Carcinoma; Nasopharyngeal Cancer; Hypothyroidism
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Nasopharyngeal Neoplasms; Hypothyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified neck target volume delineation (Experimental): For patients with negative lymph nodes in regions III and IVa, a modified neck target volume delineation method was used to define the inner boundary of regions III and IVa as the outer edge of the common carotid artery.
  Interventions: Radiation: Modified neck target volume delineation
- Routine neck target volume delineation (No Intervention): For patients with negative lymph nodes in regions III and IVa, the inner boundary of regions III and IVa is defined as the inner edge of the common carotid artery or the outer edge of the thyroid.

INTERVENTIONS:
Radiation: Modified neck target volume delineation — Modified neck target volume delineation method was used to define the inner boundary of regions III and IVa as the outer edge of the common carotid artery.
  Arms: Modified neck target volume delineation

SUMMARY:
This study aimed to reduce radiation-induced thyroid injury without compromising control of the cervical region by optimizing the delineation of the cervical lymph node drainage area.

DETAILED DESCRIPTION:
Since the neck target area of nasopharyngeal carcinoma is close to the thyroid gland, the average dose to the thyroid gland is usually around 54Gy, which is difficult to meet the protection requirements for thyroid protection. In the current guidelines, the inner edge of the common carotid artery is used as the inner boundary of the lymph nodes in levels III and IVa, and the lymphatic drainage area needs to include the inner edge of the common carotid artery. Several studies have found that the centers of positive lymph nodes in cervical regions III and IVa are located outside the inner border of the common carotid artery. In order to better protect the thyroid gland, the investigators have improved the delineation of the neck target area. For patients with negative lymph nodes in regions II and IVa (accounting for about 60% of the total patients), a modified neck target volume delineation method was used to define the inner boundary of regions III and IVa as the outer edge of the common carotid artery. For patients with positive lymph nodes in regions III and IVa (accounting for about 40% of the total patients), the inner boundary of regions III and IVa is defined as the inner edge of the common carotid artery or the outer edge of the thyroid. This study aimed to reduce radiation-induced thyroid injury without compromising control of the cervical region by optimizing the delineation of the cervical lymph node drainage area.

ELIGIBILITY:
Inclusion Criteria:

1. The pathological diagnosis was newly diagnosed non-keratinizing squamous cell carcinoma nasopharyngeal carcinoma.
2. The clinical stage is T1-4N0-3M0 (stage I~IVa, UICC/AJCC 8th edition);
3. There is no history of hypothyroidism or hyperthyroidism before treatment;
4. Using intensity-modulated radiotherapy technology,
5. Complete radical dose radiotherapy;
6. KPS≥70 points;
7. Age 18-70 years old;
8. Male or female who is not pregnant or lactating;
9. Hematological examination: white blood cells > 4×109/L, neutrophils > 2×109/L, hemoglobin > 90g/L, platelets > 100×109/L;
10. Liver function: ALT, AST < 1.5×ULN, ALP < 2.5×ULN, bilirubin < ULN.
11. Renal function: creatinine > 60 ml/min;
12. The patient signs the informed consent form;

Exclusion Criteria:

1. WHO pathological classification is keratinizing squamous cell carcinoma or basaloid carcinoma;
2. palliative treatment;
3. Have a history of other malignant tumors;
4. Pregnant or lactating women (women of childbearing age should consider taking a pregnancy test, and patients are required to use effective contraception during treatment);
5. Have a history of neck surgery;
6. Have a history of hyperthyroidism or hypothyroidism.
7. Previous history of head and neck radiation therapy;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Regional Recurrence-free Survival | 3 years
  From the date of diagnosis to the day of date of diagnosis and the date of regional relapse

SECONDARY OUTCOMES:
Radiation-induced hypothyroidism | 3 years
  From the date of diagnosis to the day of date of diagnosis and the date of regional TSH > upper limit of normal, FT4 normal or less than < lower limit of normal
Overall Survival | 3 years
  From the date of diagnosis to any death, with patients unavailable for follow-up censored at the date of last follow-up
Progression-free Survival | 3 years
  From the date of diagnosis to the data of tumor progression or death (for any cause)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nasopharyngeal Carcinoma, Jiangxi Cancer Hospital, Nanchang, None Selected, China